CLINICAL TRIAL: NCT05377723
Title: Abdominal Scar Improvement in Microsurgical Breast Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Neodyne Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-59506; NCI-2023-03670 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cicatrix; Breast Reconstruction
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Neodyne Device (Experimental): After eligible patients have provided informed consent, the side of the abdomen to be treated with the Neodyne Device will be randomly selected by opening a sealed randomization envelope. The selected side will be treated with the Neodyne Device through the full study. The Neodyne Device will be applied to a portion of the abdominal incision by the health care provider at 1 week (4-8 days) after the procedure. The other portion of the abdominal incision (Arm Title: Control) will serve as the control and will be treated per the investigator's standard of care. Subjects will return to the Investigator's office for a total of 8 weeks for application and removal of the Neodyne Dressing.
  Interventions: Device: Neodyne Device
- Control (Other): See above
  Interventions: Device: Neodyne Device

INTERVENTIONS:
Device: Neodyne Device — See Arm Description: Neodyne Device

SUMMARY:
Microsurgical breast reconstruction is most commonly performed with free abdominal flaps, which leave a long transverse lower abdominal scar. Due to tension across the incision, these scars frequently widen and hypertrophy. Hence, modalities that can reduce this tendency, thus, improving scar appearance are desirable. Here, we wish to investigate the impact of the Neodyne embrace device on postoperative abdominal scar appearance. The proposed study is novel in that it is the first RCT investigating the effect of the embrace device on scar appearance in the context of microsurgical breast reconstruction.

DETAILED DESCRIPTION:
Adult (>18 years) women who have undergone microsurgical breast reconstruction with free abdominal flap(s) approximately 1 week (5-10 days) prior to study participation will be approached by the clinical research team during their first postoperative clinic visit; the protocol asks for the device to be applied at this point. Investigators will only invite those subjects to participate whose incisions, at the 1 week postoperative visit, appear to be uniformly aesthetically similar across the length of the incision. Informed consent for randomization and study participation will be obtained.

After eligible patients have provided informed consent, the side of the abdomen to be treated with the Neodyne Device will be randomly selected by opening a sealed randomization envelope. The selected side will be treated with the Neodyne Device through the full study. The Neodyne Device will be applied to a portion of the abdominal incision by the health care provider at 1 week (4-8 days) after the procedure. The other portion of the abdominal incision will serve as the control and will be treated per the investigator's standard of care. Subjects will return to the Investigator's office for a total of 8 weeks for application and removal of the Neodyne Dressing.

At the 8th week visit subjects and investigators will complete an evaluation of the incision/scar. Subjects will return to the Investigator's office at 12 weeks from the date of the procedure for another evaluation of the incision/scar. The primary study endpoint will be evaluated at 6 months from the date of the procedure. Subjects will also be offered the opportunity to provide additional photographic evaluations at 12 months after surgery in conjunction with a standard clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. Female Subjects who have undergone unilateral/bilateral microsurgical breast reconstruction with free abdominal flaps within approximately 1 week (4-8 days) prior to study participation.
2. Appearance of subject's incision is aesthetically similar across length of incision
3. Age >18
4. Subject has the ability to read and comprehend as required by the protocol and the informed consent.
5. Subject must be able to provide written informed consent prior to participation in the study.

Exclusion Criteria:

1. Subjects with a history of collagen vascular disease, cutis laxica, connective tissue disease, psoriasis, or lupus.
2. Subjects diagnosed with scleroderma.
3. Subjects with known adverse reactions to steri-strip tapes, medical tapes, or adhesives.
4. Subjects with oozing, dehiscence, non-closed/healed incisions at time of first application.
5. Subjects with inability to maintain adequate care of incision.
6. Subjects with a weight loss of > 100 lbs within 6 months from date of surgery.
7. Subjects who currently smoke.
8. Subjects taking steroid therapy (systemic or inhaled) within 2 months from date of study enrollment.
9. Subject does not qualify for the study in the opinion of the investigators.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Scar Assessment | 6 months
  The primary endpoint is the difference between the assessments of the scar appearance for the treated as compared to the control incision sites. Incisions will be evaluated by an objective independent expert panel at six months post surgery. The panel will review close-up photographic records, taken at the 6 month study endpoint, of the control incision site and the treated incision site. The subject will complete the Scar Q questionnaire and both the investigator and the subject will complete the Patient and Observer Scar Assessment Scale (POSAS). It is expected that the scar from the incision area covered by Neodyne Dressing will be minimized when compared to the scar from the untreated incision area.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Momeni, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No